CLINICAL TRIAL: NCT06631508
Title: Development of Perioperative Follow-up Protocols and Evaluation of Their Effectiveness for Women Aged 30-65 Having Pelvic Organ Prolapse Surgery
Brief Title: Perioperative Follow-up Protocols for Pelvic Organ Prolapse Surgery
Acronym: POPFollowup
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Nazlı Özbek, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: nozbek
Record Dates: First submitted 2023-10-16; First posted 2024-10-08 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; perioperative care; follow up protocol; nursing care
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Preoperative Period; Postoperative Period

STUDY DESIGN:
Intervention Model Description: randomized controlled intervention trial After informed voluntary consent is obtained, full randomization technique will be used to assign participants to follow-up and control groups. Full randomization will be done via the website http://www.randomizer.org/. Two computer-generated randomization sequences will be applied on a one-to-one basis.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Preoperative Period, Education video (Experimental): Follow-up Group: Preoperative data of patients who will undergo pelvic organ prolapse surgery will be collected. Then, the preoperative patient education video will be watched. If patient has any questions will be answered.
  Control Group: No intervention. Control Group's data will be collected.
  Data collection forms to be used in the preoperative period:
  * Introductory Characteristics Form
  * Pelvic Organ Prolapse Quality of Life Scale
  * Pelvic Organ Prolapse Symptom Score
  * Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire
  * State-Trait Anxiety Inventory Short Version
  * Preoperative Functional Health Patterns Evaluation Form
  Interventions: Other: Preoperative Period, Postoperative Period, 2th week after discharge, 6th week after discharge, 10th week after discharge, 14th week after discharge
- Postoperative Period, Education video (Experimental): Patient data will be collected within 24-48 hours in the postoperative period. The postoperative patient education video will be watched before the patient is discharged. If patient has any questions, they will be answered.
  Control Group: No intervention. Control Group's data will be collected.
  Data collection forms to be used in the postoperative period:
  * Postoperative Data Collection Form
  * State-Trait Anxiety Inventory Short Version
  * Postoperative Functional Health Patterns Evaluation Form
  * Nursing Diagnoses Checklist After POP Surgery
  Interventions: Other: Preoperative Period, Postoperative Period, 2th week after discharge, 6th week after discharge, 10th week after discharge, 14th week after discharge
- 2th week after discharge (Experimental): The patient's data will be collected by telephone follow-up two weeks after discharge.
  Control Group: No intervention. Control Group's data will be collected.
  Data collection forms to be used at the two weeks after discharge:
  * Pelvic Organ Prolapse Quality of Life Scale
  * Pelvic Organ Prolapse Symptom Score
  * State-Trait Anxiety Inventory Short Version
  * After Discharge Functional Health Patterns Evaluation Form
  * Nursing Diagnoses Checklist After POP Surgery
  Interventions: Other: Preoperative Period, Postoperative Period, 2th week after discharge, 6th week after discharge, 10th week after discharge, 14th week after discharge
- 6th week after discharge (Experimental): The patient's data will be collected by telephone follow-up six weeks after discharge.
  Control Group: No intervention. Control Group's data will be collected.
  Data collection forms to be used at the six weeks after discharge:
  * Pelvic Organ Prolapse Quality of Life Scale
  * Pelvic Organ Prolapse Symptom Score
  * State-Trait Anxiety Inventory Short Version
  * After Discharge Functional Health Patterns Evaluation Form
  * Nursing Diagnoses Checklist After POP Surgery
  Interventions: Other: Preoperative Period, Postoperative Period, 2th week after discharge, 6th week after discharge, 10th week after discharge, 14th week after discharge
- 10th week after discharge (Experimental): The patient's data will be collected by telephone follow-up ten weeks after discharge.
  Control Group: No intervention. Control Group's data will be collected.
  Data collection forms to be used at the ten weeks after discharge:
  * Pelvic Organ Prolapse Quality of Life Scale
  * Pelvic Organ Prolapse Symptom Score
  * State-Trait Anxiety Inventory Short Version
  * After Discharge Functional Health Patterns Evaluation Form
  * Nursing Diagnoses Checklist After POP Surgery
  Interventions: Other: Preoperative Period, Postoperative Period, 2th week after discharge, 6th week after discharge, 10th week after discharge, 14th week after discharge
- 14th week after discharge (Experimental): The patient's data will be collected by telephone follow-up fourteen weeks after discharge. Additionally, on the 14th week, a satisfaction form will be applied to the Follow-up Group to evaluate the education videos.
  Control Group: No intervention. Control Group's data will be collected. After the data is collected, postoperative education video will be watched.
  Data collection forms to be used at the fourteen weeks after discharge:
  * Pelvic Organ Prolapse Quality of Life Scale
  * Pelvic Organ Prolapse Symptom Score
  * Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire
  * State-Trait Anxiety Inventory Short Version
  * After Discharge Functional Health Patterns Evaluation Form
  * Nursing Diagnoses Checklist After POP Surgery
  * Satisfaction Evaluation Form (Only Follow-up Group)
  Interventions: Other: Preoperative Period, Postoperative Period, 2th week after discharge, 6th week after discharge, 10th week after discharge, 14th week after discharge

INTERVENTIONS:
Other: Preoperative Period, Postoperative Period, 2th week after discharge, 6th week after discharge, 10th week after discharge, 14th week after discharge — Showing training videos to patients before and after pelvic organ prolapse surgery and following up after discharge

SUMMARY:
The goal of this clinical trial is to develop perioperative follow-up and evaluation of their effectiveness protocols in women aged 30-65 having pelvic organ prolapse surgery.

The main questions it aims to answer are:

* Is the perioperative follow up protocol developed for women aged 30-65 having pelvic organ prolapse surgery effective?
* Does the developed perioperative follow up protocol for women aged 30-65 having pelvic organ prolapse surgery have an effect on quality of life, pelvic organ symptom score, sexual function, functional health patterns and anxiety?

DETAILED DESCRIPTION:
In order to maintain holistic care, maintaining communication with the individual after discharge and providing individual counseling regarding the problems experienced have an important place in patient follow-up. In this context, perioperative consultancy should be provided under nurse management to make it easier for patients to cope with physical and psychosocial problems, improve quality of life and ensure continuity of care. Therefore, in this research; the aim is to develop perioperative follow up protocols and evaluate their effectiveness for women aged 30-65 who have pelvic organ prolapse surgery.

The sample of the research; It is planned to consist of a total of 102 women, 51 in the Follow-up Group and 51 in the Control Group, who meet the inclusion criteria and voluntarily agreed to participate in the research (Calculated using G.Power 3.1.7 program). After informed consent is obtained, full randomization technique will be used to assign participants to follow-up and control groups. Full randomization will be done via the website http://www.randomizer.org/. Two computer-generated randomization sequences will be applied on a one-to-one basis.

During the pre-test and post-test data collection phase, it is planned to use the 'Descriptive Characteristics Form', 'Pelvic Organ Prolapse Quality of Life Scale', 'Pelvic Organ Symptom Score', 'Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire Form', 'State-Trait Anxiety Inventory Short Version', and 'Functional Health Patterns Assessment Form' in the perioperative period.

After preoperative data is collected, the Follow-up Group will be shown a preoperative patient education video. In the postoperative period, Follow-up Group's data will be collected within 24-48 hours and the patient will be shown a postoperative education video before discharge. After discharge; at the 2nd, 6th, 10th and 14th weeks, Follow-up Group's will be followed up by phone and their data will be collected. In addition, a satisfaction form to evaluate the education videos will be applied to the Follow-up Group in the 14th week. The Control Group will not receive any intervention by the researcher and will receive routine perioperative care. Control Group's data will be collected in the preoperative and postoperative period. Additionally, Control Group's data will be collected by phone at the 2nd, 6th, 10th and 14th weeks after discharge and a postoperative education video will be watched after the data is collected at the 14th week.

ELIGIBILITY:
Inclusion Criteria:

* Being stage ≥2 according to POP Classification (POP-Q),
* Being between 30-65 years old,
* Being sexually active,
* Ability to read and write,
* Ability to speak Turkish,
* Ability to use phone
* Having a phone that can be reached at all times and
* Agreeing to participate in the study

Exclusion Criteria:

* Being stage <2 according to POP Classification (POP-Q),
* Being between <30 and >65 years of age,
* Not being sexually active,
* Not being able to read and write,
* Not being able to speak Turkish,
* Inability to use the phone
* Not having a phone that can be reached at all times and
* Not agreeing to participate in the study
* Discontinue the research for any reason

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Scale | Baseline and at 2, 6, 10 and 14 weeks postoperatively
  Evaluation of the quality of life of women who had pelvic organ prolapse surgery before and after the study.
  The scale was developed to evaluate the general health perceptions of patients with pelvic organ prolapse, the symptoms experienced during prolapse, and the effects and consequences of symptoms on quality of life. The scale consists of eight areas. There is no total score for the areas used in the scale, each area is scored individually.In calculating the score of the areas; a four-point scoring system is used for the expressions; does not affect at all, slightly affects, moderately affects and greatly affects; 1, 2, 3, 4, respectively. Each area of the scale is calculated separately depending on the questions it contains. The scale is scored between 0 and 100. High scores obtained from the scale indicate that the quality of life is impaired, while low scores indicate that the quality of life is better.
Functional Health Patterns | Baseline and at 24.-48hours and 2, 6, 10 and 14 weeks postoperatively.
  Evaluation of the health patterns of women who had pelvic organ prolapse surgery before and after study.
  It was developed by researchers in line with the relevant literature according to Gordon's Functional Health Patterns. The form, which is created separately for the preoperative, postoperative and post-discharge periods, covers 11 areas such as health perception, nutrition, excretion, activity, sleep, cognitive-perception style. The preoperative, postoperative and post-discharge health status of the patients, the problems they experience and the complications that may develop are determined. The items in the form are evaluated with yes-no and 0-10 (0 not affected at all, 10 affected a lot) Visual Analog Scale (VAS) and 5-point Likert (very good - good - medium - bad - very bad). There is no total score from the form. Each question is evaluated on its own.

SECONDARY OUTCOMES:
Pelvic Organ Symptom Score | Baseline and at 2, 6, 10 and 14 weeks postoperatively.
  Evaluation of the pelvic organ symptom score of women who had pelvic organ prolapse surgery before and after study. The scale is used to evaluate symptoms of pelvic organ prolapse. There are seven questions in the scale, each with five answers. The answers are formed as never (0 points), a little (1 point), sometimes (2 points), often (3 points) and always (4 points). An increase in the score obtained from the scale indicates an increase in symptoms. In addition, women indicate which of the seven symptoms bother them the most.
Sexual Function | Baseline and after 14 weeks
  Evaluation of sexual function of women who had pelvic organ prolapse surgery before and after study. Questionnaire developed to evaluate sexual function specific to the urogynecological field consists of 12 items. Questions 1-4 on the form are scored as 4 points = always and 0 = never, while questions 5-12 are scored as 0 = always and 4 points = never. A minimum of 0 and a maximum of 48 points can be obtained from the questionnaire. As the score of the questionnaire increases, it indicates an improvement in sexual function. The questionnaire is divided into three sub-dimensions: behavioral/emotional status (questions 1-4), physical status (questions 5-9) and partner-related status (questions 10-12).
Anxiety | Baseline and at 2, 6, 10 and 14 weeks postoperatively.
  Evaluation of the anxiety of women who had pelvic organ prolapse surgery before and after study. Two scales measuring state and trait anxiety are used. The scales consist of 5 items and are of 4-point Likert type. Individuals who score 10 and above on State Anxiety Inventory Scale-5 and 14 and above on Trait Anxiety Inventory Scale-5 are considered to be clinically anxious.
Nursing Diagnosis Checklist | At 2, 6, 10 and 14 weeks postoperatively.
  This form prepared by researchers lists nursing diagnoses to identify problems that may develop in patients at 24-48 hours postoperatively and at 2, 6, 10 and 14 weeks after discharge. These diagnoses are systematized in 11 areas according to Gordon's Functional Health Patterns Model. There is no score calculation in this form, and the most frequently used diagnoses will be calculated as percentages.
Satisfaction Evaluation Form | At 14 weeks postoperatively.
  This form, developed by the researchers, will be applied to the follow-up group in the 14th week. This form will determine the patients' satisfaction levels regarding the preoperative and postoperative education videos. The form, consisting of 12 items, is evaluated with a 5-point Likert scale (Not satisfied at all = 0 points, not satisfied = 1 point, undecided = 2 points, satisfied = 3 points, very satisfied = 4 points). As the score increases, satisfaction increases.

CONTACTS AND LOCATIONS:
Overall Officials: Gulsah Kök, Study Director — SBU Health Science Faculty Gulhane Nursing Faculty
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Hendrix SL, Clark A, Nygaard I, Aragaki A, Barnabei V, McTiernan A. Pelvic organ prolapse in the Women's Health Initiative: gravity and gravidity. Am J Obstet Gynecol. 2002 Jun;186(6):1160-6. doi: 10.1067/mob.2002.123819. PMID 12066091
- [Background] Weintraub AY, Glinter H, Marcus-Braun N. Narrative review of the epidemiology, diagnosis and pathophysiology of pelvic organ prolapse. Int Braz J Urol. 2020 Jan-Feb;46(1):5-14. doi: 10.1590/S1677-5538.IBJU.2018.0581. PMID 31851453
- [Background] Rogers RG, Coates KW, Kammerer-Doak D, Khalsa S, Qualls C. A short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). Int Urogynecol J Pelvic Floor Dysfunct. 2003 Aug;14(3):164-8; discussion 168. doi: 10.1007/s00192-003-1063-2. Epub 2003 Jul 25. PMID 12955337
- [Background] Hagen S, Glazener C, Sinclair L, Stark D, Bugge C. Psychometric properties of the pelvic organ prolapse symptom score. BJOG. 2009 Jan;116(1):25-31. doi: 10.1111/j.1471-0528.2008.01903.x. Epub 2008 Oct 8. PMID 18947342
- [Background] Digesu GA, Khullar V, Cardozo L, Robinson D, Salvatore S. P-QOL: a validated questionnaire to assess the symptoms and quality of life of women with urogenital prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2005 May-Jun;16(3):176-81; discussion 181. doi: 10.1007/s00192-004-1225-x. Epub 2004 Oct 21. PMID 15875234
- [Background] Zhang T, Qi X. Enhanced Nursing Care for Improving the Self-Efficacy & Health-Related Quality of Life in Patients with a Urostomy. J Multidiscip Healthc. 2023 Jan 29;16:297-308. doi: 10.2147/JMDH.S394515. eCollection 2023. PMID 36741293
- [Background] Rockefeller NF, Jeppson P, Komesu YM, Meriwether KV, Ninivaggio C, Dunivan G. Preferences for Preoperative Education: A Qualitative Study of the Patient Perspective. Female Pelvic Med Reconstr Surg. 2021 Oct 1;27(10):633-636. doi: 10.1097/SPV.0000000000001014. PMID 34554145
- [Background] Richardson K, Hagen S. The role of nurses in the management of women with pelvic organ prolapse. Br J Nurs. 2009 Mar 12-25;18(5):294-6, 298-300. doi: 10.12968/bjon.2009.18.5.40710. PMID 19374034
- [Background] Haya N, Feiner B, Baessler K, Christmann-Schmid C, Maher C. Perioperative interventions in pelvic organ prolapse surgery. Cochrane Database Syst Rev. 2018 Aug 19;8(8):CD013105. doi: 10.1002/14651858.CD013105. PMID 30121957
- [Result] Belayneh T, Gebeyehu A, Adefris M, Rortveit G, Gjerde JL, Ayele TA. Pelvic organ prolapse surgery and health-related quality of life: a follow-up study. BMC Womens Health. 2021 Jan 2;21(1):4. doi: 10.1186/s12905-020-01146-8. PMID 33388056